CLINICAL TRIAL: NCT00005132
Title: National Growth and Health Study (NGHS)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1002
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2006-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Coronary Disease; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Coronary Disease; Hypertension

SUMMARY:
To determine if the Black-white differences in the development of obesity in pubescent females were due to differences in psychosocial, socioeconomic and other environmental factors. Also, to determine whether differences in the development of obesity led to Black-white differences in other coronary heart disease risk factors, such as blood pressure and serum lipids.

DETAILED DESCRIPTION:
BACKGROUND:

Although not all scientists agree that obesity is an independent risk factor for coronary heart disease, it may be a strong univariate predictor of coronary heart disease, and impacts on coronary heart disease through at least some of its relationships with other risk factors: positive association with blood pressure, inverse association with high density lipoprotein cholesterol (HDLC), positive association with triglyceride and very low density lipoprotein cholesterol (VLDLC), and a positive association with hyperglycemia and diabetes. A number of these have been shown to be major coronary heart disease risk factors. Prevention of obesity, or weight reduction towards desirable body weight may reduce the incidence of coronary heart disease and some of its risk factors. There is evidence to suggest that once obesity begins and/or advances in childhood, it will track into adulthood, with a reasonably high level of certainty. Obesity becomes progressively more difficult to treat with maturation to adulthood. Thus, better understanding of the pathophysiology of obesity in late childhood and early adolescence should, in the long-run, provide the basis for effective prevention or intervention programs in order to have a long-range impact upon the consequence of obesity. The age group 9 and 10 at entry has been selected to assure that many of the individuals are enrolled prior to puberty, and followed through this transition period when obesity becomes more apparent among Black adolescent females than among white.

Support for this research grew out of recommendations made at the Working Conference on Coronary Heart Disease in Black Populations held in September 1983 and sponsored by the NHLBI. The group recommended this research to identify the physiological and/or behavioral factors which contribute to obesity in Black females. In addition, the 1981 Report of the Working Group on Arteriosclerosis of the NHLBI stated that research is needed to characterize the behaviors that create and maintain caloric imbalance. The initiative was approved by the September 1984 National Heart, Lung, and Blood Advisory Council and the Request for Proposals was released in November 1984.

The NGHS I was initiated in 1985 as a contract-supported program with three field centers and a coordinating center. Annual exams were conducted at baseline and through the years of follow-up. The study was renewed by means of the cooperative agreement mechanism in 1992 as the NGHS II to permit two additional years of follow-up exams. The study was again renewed in 1994 as NGHS III to continue annual examinations.

DESIGN NARRATIVE:

In this longitudinal study, there were a baseline examination and annual examinations. Data collected included: physical examination; anthropometric measurements; dietary information including food pattern and nutrient intake; physical activity; lipid, lipoprotein, and apolipoprotein profiles; family socioeconomic status; and psychosocial information. The study was renewed twice to continue the longitudinal investigation until the subjects reached the age of 19 to 20. Following the girls until that age allowed the documentation of the transition in risk factors when Black girls no longer have a cardiovascular risk advantage and to study the factors surrounding the transition. The longer follow-up also allowed for studies on the influence of smoking on body weight and the relationship of adolescent pregnancy to subsequent adiposity development, body fat patterning, blood pressure, and blood lipids.

ELIGIBILITY:
No eligibility criteria

Ages: 9 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1985-09; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barton — Maryland Medical Research Institute; Paul Canner — Maryland Medical Research Institute; Stephen Daniels — Children's Hospital & Medical Center; John Morrison — University of Cincinnati; Z.I. Sabry — University of California at Berkeley; George Schreiber — Westat, Inc.

REFERENCES:
- [Background] Schumann BC, Striegel-Moore RH, McMahon RP, Waclawiw MA, Morrison JA, Schreiber GB. Psychometric properties of the Self-Perception Profile for Children in a biracial cohort of adolescent girls: the NHLBI Growth and Health Study. J Pers Assess. 1999 Oct;73(2):260-75. doi: 10.1207/S15327752JPA7302_5. PMID 10624004
- [Background] Morrison JA, Sprecher DL, Barton BA, Waclawiw MA, Daniels SR. Overweight, fat patterning, and cardiovascular disease risk factors in black and white girls: The National Heart, Lung, and Blood Institute Growth and Health Study. J Pediatr. 1999 Oct;135(4):458-64. doi: 10.1016/s0022-3476(99)70168-x. PMID 10518079
- [Background] Kimm SY, Pasagian-Macaulay A, Aston CE, McAllister AE, Glynn NW, Kamboh MI, Ferrell RE. Correlates of lipoprotein(a) levels in a biracial cohort of young girls: the NHLBI Growth and Health Study. J Pediatr. 1999 Aug;135(2 Pt 1):169-76. doi: 10.1016/s0022-3476(99)70018-1. PMID 10431110
- [Background] Striegel-Moore RH, Morrison JA, Schreiber G, Schumann BC, Crawford PB, Obarzanek E. Emotion-induced eating and sucrose intake in children: the NHLBI Growth and Health Study. Int J Eat Disord. 1999 May;25(4):389-98. doi: 10.1002/(sici)1098-108x(199905)25:43.0.co;2-4. PMID 10202649
- [Background] Patterson ML, Stern S, Crawford PB, McMahon RP, Similo SL, Schreiber GB, Morrison JA, Waclawiw MA. Sociodemographic factors and obesity in preadolescent black and white girls: NHLBI's Growth and Health Study. J Natl Med Assoc. 1997 Sep;89(9):594-600. PMID 9302856
- [Background] Sprecher DL, Morrison JA, Simbartl LA, Schreiber GB, Sabry ZI, Biro FM, Barton BA. Lipoprotein and apolipoprotein differences in black and white girls. The National Heart, Lung, and Blood Institute Growth and Health Study. Arch Pediatr Adolesc Med. 1997 Jan;151(1):84-90. doi: 10.1001/archpedi.1997.02170380088014. PMID 9006534
- [Background] Daniels SR, Obarzanek E, Barton BA, Kimm SY, Similo SL, Morrison JA. Sexual maturation and racial differences in blood pressure in girls: the National Heart, Lung, and Blood Institute Growth and Health Study. J Pediatr. 1996 Aug;129(2):208-13. doi: 10.1016/s0022-3476(96)70244-5. PMID 8765617
- [Background] Kimm SY, Obarzanek E, Barton BA, Aston CE, Similo SL, Morrison JA, Sabry ZI, Schreiber GB, McMahon RP. Race, socioeconomic status, and obesity in 9- to 10-year-old girls: the NHLBI Growth and Health Study. Ann Epidemiol. 1996 Jul;6(4):266-75. doi: 10.1016/s1047-2797(96)00056-7. PMID 8876836
- [Background] Schreiber GB, Robins M, Striegel-Moore R, Obarzanek E, Morrison JA, Wright DJ. Weight modification efforts reported by black and white preadolescent girls: National Heart, Lung, and Blood Institute Growth and Health Study. Pediatrics. 1996 Jul;98(1):63-70. PMID 8668414
- [Background] Morrison JA, Sprecher D, McMahon RP, Simon J, Schreiber GB, Khoury PR. Obesity and high-density lipoprotein cholesterol in black and white 9- and 10-year-old girls: The National Heart, Lung, and Blood Institute Growth and Health Study. Metabolism. 1996 Apr;45(4):469-74. doi: 10.1016/s0026-0495(96)90221-8. PMID 8609833
- [Background] Biro FM, Daniels SR, Similo SL, Barton BA, Payne GH, Morrison JA. Differential classification of blood pressure by fourth and fifth Korotkoff phases in school-aged girls. The National Heart, Lung, and Blood Institute Growth and Health Study. Am J Hypertens. 1996 Mar;9(3):242-7. doi: 10.1016/0895-7061(95)00295-2. PMID 8695023
- [Background] Crawford PB, Obarzanek E, Schreiber GB, Barrier P, Goldman S, Frederick MM, Sabry ZI. The effects of race, household income, and parental education on nutrient intakes of 9- and 10-year-old girls. NHLBI Growth and Health Study. Ann Epidemiol. 1995 Sep;5(5):360-8. doi: 10.1016/1047-2797(95)00033-4. PMID 8653208
- [Background] Obarzanek E, Schreiber GB, Crawford PB, Goldman SR, Barrier PM, Frederick MM, Lakatos E. Energy intake and physical activity in relation to indexes of body fat: the National Heart, Lung, and Blood Institute Growth and Health Study. Am J Clin Nutr. 1994 Jul;60(1):15-22. doi: 10.1093/ajcn/60.1.15. PMID 8017331
- [Background] Morrison JA, Barton B, Biro FM, Sprecher DL, Falkner F, Obarzanek E. Sexual maturation and obesity in 9- and 10-year-old black and white girls: the National Heart, Lung, and Blood Institute Growth and Health Study. J Pediatr. 1994 Jun;124(6):889-95. doi: 10.1016/s0022-3476(05)83176-2. PMID 8201472
- [Background] Crawford PB, Obarzanek E, Morrison J, Sabry ZI. Comparative advantage of 3-day food records over 24-hour recall and 5-day food frequency validated by observation of 9- and 10-year-old girls. J Am Diet Assoc. 1994 Jun;94(6):626-30. doi: 10.1016/0002-8223(94)90158-9. PMID 8195550
- [Background] Campaigne BN, Morrison JA, Schumann BC, Falkner F, Lakatos E, Sprecher D, Schreiber GB. Indexes of obesity and comparisons with previous national survey data in 9- and 10-year-old black and white girls: the National Heart, Lung, and Blood Institute Growth and Health Study. J Pediatr. 1994 May;124(5 Pt 1):675-80. doi: 10.1016/s0022-3476(05)81354-x. PMID 8176552
- [Background] Simon JA, Obarzanek E, Daniels SR, Frederick MM. Dietary cation intake and blood pressure in black girls and white girls. Am J Epidemiol. 1994 Jan 15;139(2):130-40. doi: 10.1093/oxfordjournals.aje.a116975. PMID 8296780
- [Background] Simon JA, Schreiber GB, Crawford PB, Frederick MM, Sabry ZI. Income and racial patterns of dietary vitamin C intake among black and white girls. Public Health Rep. 1993 Nov-Dec;108(6):760-4. PMID 8265761
- [Background] Obesity and cardiovascular disease risk factors in black and white girls: the NHLBI Growth and Health Study. Am J Public Health. 1992 Dec;82(12):1613-20. doi: 10.2105/ajph.82.12.1613. PMID 1456335
- [Background] Brown KM, McMahon RP, Biro FM, Crawford P, Schreiber GB, Similo SL, Waclawiw M, Striegel-Moore R. Changes in self-esteem in black and white girls between the ages of 9 and 14 years. The NHLBI Growth and Health Study. J Adolesc Health. 1998 Jul;23(1):7-19. doi: 10.1016/s1054-139x(97)00238-3. PMID 9648018
- [Background] Kimm SY, Barton BA, Berhane K, Ross JW, Payne GH, Schreiber GB. Self-esteem and adiposity in black and white girls: the NHLBI Growth and Health Study. Ann Epidemiol. 1997 Nov;7(8):550-60. doi: 10.1016/s1047-2797(97)00124-5. PMID 9408551
- [Background] McNutt SW, Hu Y, Schreiber GB, Crawford PB, Obarzanek E, Mellin L. A longitudinal study of the dietary practices of black and white girls 9 and 10 years old at enrollment: the NHLBI Growth and Health Study. J Adolesc Health. 1997 Jan;20(1):27-37. doi: 10.1016/S1054-139X(96)00176-0. PMID 9007656
- [Background] Simon JA, Morrison JA, Similo SL, McMahon RP, Schreiber GB. Correlates of high-density lipoprotein cholesterol in Black girls and White girls: the NHLBI Growth and Health Study. Am J Public Health. 1995 Dec;85(12):1698-702. doi: 10.2105/ajph.85.12.1698. PMID 7503349
- [Background] Striegel-Moore RH, Schreiber GB, Pike KM, Wilfley DE, Rodin J. Drive for thinness in black and white preadolescent girls. Int J Eat Disord. 1995 Jul;18(1):59-69. doi: 10.1002/1098-108x(199507)18:13.0.co;2-6. PMID 7670444
- [Background] Morrison JA, Payne G, Barton BA, Khoury PR, Crawford P. Mother-daughter correlations of obesity and cardiovascular disease risk factors in black and white households: the NHLBI Growth and Health Study. Am J Public Health. 1994 Nov;84(11):1761-7. doi: 10.2105/ajph.84.11.1761. PMID 7977914
- [Background] Wang MC, Moore EC, Crawford PB, Hudes M, Sabry ZI, Marcus R, Bachrach LK. Influence of pre-adolescent diet on quantitative ultrasound measurements of the calcaneus in young adult women. Osteoporos Int. 1999;9(6):532-5. doi: 10.1007/s001980050181. PMID 10624461
- [Background] Simon JA, Schreiber GB, Crawford PB, Frederick MM, Sabry ZI. Dietary vitamin C and serum lipids in black and white girls. Epidemiology. 1993 Nov;4(6):537-42. doi: 10.1097/00001648-199311000-00010. PMID 8268283
- [Background] Daniels SR, McMahon RP, Obarzanek E, Waclawiw MA, Similo SL, Biro FM, Schreiber GB, Kimm SY, Morrison JA, Barton BA. Longitudinal correlates of change in blood pressure in adolescent girls. Hypertension. 1998 Jan;31(1):97-103. doi: 10.1161/01.hyp.31.1.97. PMID 9449398
- [Background] Striegel-Moore RH, Schreiber GB, Lo A, Crawford P, Obarzanek E, Rodin J. Eating disorder symptoms in a cohort of 11 to 16-year-old black and white girls: the NHLBI growth and health study. Int J Eat Disord. 2000 Jan;27(1):49-66. doi: 10.1002/(sici)1098-108x(200001)27:13.0.co;2-e. PMID 10590449
- [Background] Morrison JA, Barton BA, Obarzanek E, Crawford PB, Guo SS, Schreiber GB, Waclawiw M. Racial differences in the sums of skinfolds and percentage of body fat estimated from impedance in black and white girls, 9 to 19 years of age: the National Heart, Lung, and Blood Institute Growth and Health Study. Obes Res. 2001 May;9(5):297-305. doi: 10.1038/oby.2001.37. PMID 11346671
- [Background] Biro FM, McMahon RP, Striegel-Moore R, Crawford PB, Obarzanek E, Morrison JA, Barton BA, Falkner F. Impact of timing of pubertal maturation on growth in black and white female adolescents: The National Heart, Lung, and Blood Institute Growth and Health Study. J Pediatr. 2001 May;138(5):636-43. doi: 10.1067/mpd.2001.114476. PMID 11343036
- [Background] Kimm SY, Barton BA, Obarzanek E, McMahon RP, Sabry ZI, Waclawiw MA, Schreiber GB, Morrison JA, Similo S, Daniels SR. Racial divergence in adiposity during adolescence: The NHLBI Growth and Health Study. Pediatrics. 2001 Mar;107(3):E34. doi: 10.1542/peds.107.3.e34. PMID 11230615
- [Background] Wu Y, Schreiber GB, Klementowicz V, Biro F, Wright D. Racial differences in accuracy of self-assessment of sexual maturation among young black and white girls. J Adolesc Health. 2001 Mar;28(3):197-203. doi: 10.1016/s1054-139x(00)00163-4. PMID 11226842
- [Background] Voorhees CC, Schreiber GB, Schumann BC, Biro F, Crawford PB. Early predictors of daily smoking in young women: the national heart, lung, and blood institute growth and health study. Prev Med. 2002 Jun;34(6):616-24. doi: 10.1006/pmed.2002.1026. PMID 12052022
- [Background] Kimm SY, Glynn NW, Kriska AM, Barton BA, Kronsberg SS, Daniels SR, Crawford PB, Sabry ZI, Liu K. Decline in physical activity in black girls and white girls during adolescence. N Engl J Med. 2002 Sep 5;347(10):709-15. doi: 10.1056/NEJMoa003277. PMID 12213941
- [Background] Klein DJ, Aronson Friedman L, Harlan WR, Barton BA, Schreiber GB, Cohen RM, Harlan LC, Morrison JA. Obesity and the development of insulin resistance and impaired fasting glucose in black and white adolescent girls: a longitudinal study. Diabetes Care. 2004 Feb;27(2):378-83. doi: 10.2337/diacare.27.2.378. PMID 14747217
- [Background] Schmidt M, Affenito SG, Striegel-Moore R, Khoury PR, Barton B, Crawford P, Kronsberg S, Schreiber G, Obarzanek E, Daniels S. Fast-food intake and diet quality in black and white girls: the National Heart, Lung, and Blood Institute Growth and Health Study. Arch Pediatr Adolesc Med. 2005 Jul;159(7):626-31. doi: 10.1001/archpedi.159.7.626. PMID 15996994
- [Background] Affenito SG, Thompson DR, Barton BA, Franko DL, Daniels SR, Obarzanek E, Schreiber GB, Striegel-Moore RH. Breakfast consumption by African-American and white adolescent girls correlates positively with calcium and fiber intake and negatively with body mass index. J Am Diet Assoc. 2005 Jun;105(6):938-45. doi: 10.1016/j.jada.2005.03.003. PMID 15942545
- [Background] Franko DL, Thompson D, Barton BA, Dohm FA, Kraemer HC, Iachan R, Crawford PB, Schreiber GB, Daniels SR, Striegel-Moore RH. Prevalence and comorbidity of major depressive disorder in young black and white women. J Psychiatr Res. 2005 May;39(3):275-83. doi: 10.1016/j.jpsychires.2004.08.010. PMID 15725426
- [Background] Kimm SY, Glynn NW, Obarzanek E, Kriska AM, Daniels SR, Barton BA, Liu K. Relation between the changes in physical activity and body-mass index during adolescence: a multicentre longitudinal study. Lancet. 2005 Jul 23-29;366(9482):301-7. doi: 10.1016/S0140-6736(05)66837-7. PMID 16039332
- [Background] Barton BA, Eldridge AL, Thompson D, Affenito SG, Striegel-Moore RH, Franko DL, Albertson AM, Crockett SJ. The relationship of breakfast and cereal consumption to nutrient intake and body mass index: the National Heart, Lung, and Blood Institute Growth and Health Study. J Am Diet Assoc. 2005 Sep;105(9):1383-9. doi: 10.1016/j.jada.2005.06.003. PMID 16129079
- [Background] Franko DL, Striegel-Moore RH, Thompson D, Schreiber GB, Daniels SR. Does adolescent depression predict obesity in black and white young adult women? Psychol Med. 2005 Oct;35(10):1505-13. doi: 10.1017/S0033291705005386. PMID 16164774
- [Background] Morrison JA, Friedman LA, Harlan WR, Harlan LC, Barton BA, Schreiber GB, Klein DJ. Development of the metabolic syndrome in black and white adolescent girls: a longitudinal assessment. Pediatrics. 2005 Nov;116(5):1178-82. doi: 10.1542/peds.2004-2358. PMID 16264006
- [Background] Striegel-Moore RH, Thompson DR, Affenito SG, Franko DL, Barton BA, Schreiber GB, Daniels SR, Schmidt M, Crawford PB. Fruit and vegetable intake: Few adolescent girls meet national guidelines. Prev Med. 2006 Mar;42(3):223-8. doi: 10.1016/j.ypmed.2005.11.018. Epub 2006 Jan 10. PMID 16406116
- [Background] Franko DL, Thompson D, Russell R, Schreiber GB, Crawford PB, Daniels SR, Striegel-Moore RH. Correlates of persistent thinness in black and white young women. Obes Res. 2005 Nov;13(11):2006-13. doi: 10.1038/oby.2005.246. PMID 16339133
- [Background] Franko DL, Striegel-Moore RH, Bean J, Barton BA, Biro F, Kraemer HC, Schreiber GB, Crawford PB, Daniels SR. Self-reported symptoms of depression in late adolescence to early adulthood: a comparison of African-American and Caucasian females. J Adolesc Health. 2005 Dec;37(6):526-9. doi: 10.1016/j.jadohealth.2004.08.028. PMID 16310134
- [Background] Franko DL, Striegel-Moore RH, Bean J, Tamer R, Kraemer HC, Dohm FA, Crawford PB, Schreiber G, Daniels SR. Psychosocial and health consequences of adolescent depression in Black and White young adult women. Health Psychol. 2005 Nov;24(6):586-93. doi: 10.1037/0278-6133.24.6.586. PMID 16287404
- [Background] Striegel-Moore RH, Franko DL, Thompson D, Barton B, Schreiber GB, Daniels SR. Caffeine intake in eating disorders. Int J Eat Disord. 2006 Mar;39(2):162-5. doi: 10.1002/eat.20216. PMID 16231346
- [Derived] Laraia B, Brownell K, Friebur R, Perera R, Brown E, Mayer SE, Feng I, Clermont S, Ritchie LD, Epel E. Cohort profile: the longitudinal National Growth and Health Study (NGHS) of black and white girls from Northern California tracking how behavioural and psychosocial risk factors predict cardiovascular risk and biological ageing in midlife and in offspring. BMJ Open. 2023 Nov 6;13(11):e072957. doi: 10.1136/bmjopen-2023-072957. PMID 37931968
- Available data/document: Individual Participant Data Set: NGHS — http://biolincc.nhlbi.nih.gov/studies/nghs/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/nghs/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/nghs/